CLINICAL TRIAL: NCT05433948
Title: Diagnostik Af Minimal Hepatisk Encephalopati: Association Mellem Kontinuert Reaktionsstidsmåling Og EEG-indices
Brief Title: Diagnosing Minimal Hepatic Encephalopathy
Acronym: MindTheLiver
Status: Enrolling by invitation | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Regionshospitalet Silkeborg (Other); Herlev Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mette Munk Lauridsen, Associate professor, University of Southern Denmark
Other Study IDs: S-20180127
Record Dates: First submitted 2022-06-12; First posted 2022-06-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Encephalopathy; Liver Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A biobank will be set up containing blood, urine, saliva, and feces from the project participants, incl. the healthy control persons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Liver cirrhosis with normal cognition: Liver cirrhosis and performs normally in all psychometric tests. n=100
  Interventions: Diagnostic Test: Simultaneous EEG and CRT
- Liver cirrhosis with minimal hepatic encephalopathy: Liver cirrhosis and performs abnormally en 2 or more psychometric test. n=100
  Interventions: Diagnostic Test: Simultaneous EEG and CRT
- Liver cirrhosis and overt hepatic encephalopathy: West Haven grade 2 or more. n=50
  Interventions: Diagnostic Test: Simultaneous EEG and CRT
- Healthy control persons: Completely healthy persons, age, and gender-matched to cirrhosis patients. n=100
  Interventions: Diagnostic Test: Simultaneous EEG and CRT
- Sick control persons: Persons with other chronic diseases than liver disease. n=100
  Interventions: Diagnostic Test: Simultaneous EEG and CRT
- Pre-cirrhotic liver disease: Not yet cirrhosis. Will primarily be NAFLD patients. n=100
  Interventions: Diagnostic Test: Simultaneous EEG and CRT

INTERVENTIONS:
Diagnostic Test: Simultaneous EEG and CRT — EEG is recorded with 32 electrodes and commercial recording equipment.10 min EEG is recorded in idle mode with eyes closed prior to continuous EEG recording during the CRT examination, see below.
  The test is performed via a laptop using EKHO software. The software generates 150 sound stimuli of 90 dB, which the patient hears in sound-insulated headphones. Via a push button in the dominant hand, the patient must respond as quickly as possible as soon as sounds are perceived.
  PSE test: Duration 20 min. Includes 5 tasks: Digit-symbol Test, Number Connecting Test A, Number Connecting Test B, Serial Dotting Test and Line Tracing Test. Exits in 4 versions, which are used in repeated tests to avoid the learning effect. Scores range from -18 t0 6 and less -4 is abnormal.
  Other Names: PSE test; Animal Naming Test

SUMMARY:
Our purpose is to

1. Examine the correlation between MDF in a resting EEG, recorded just before the CRT test, and the variance in reaction times indicated by the CRT index
2. At simultaneous CRT and EEG recording, examine whether a change in EEG is seen immediately before an extended reaction time occurs (defined by the 75th percentile). This will shed light on a direct pathophysiological association between what is measured with EEG and CRT.
3. Investigate whether cyclicity can be detected in the continuous reaction times and if so, whether amplitude and wavelength in this cyclic activity are correlated to EEG parameters.
4. Examine whether a response to standard HE treatment can be detected with EEG in patients who are thought to suffer from it. As well as if baseline outcome predict future hepatic encephalopathy.
5. With a view to further validating our findings, investigators want to correlate results from EEG and CRT with the most internationally widespread psychometric test, the Portosystemic Encephalopathy test (PSE), which necessitates the establishment of Danish normal values. A secondary purpose of this study is therefore
6. To establish Danish normal values for the PSE test and the Animal Naming test in Danes

ELIGIBILITY:
Inclusion criteria for patients with liver cirrhosis:

1. Age> 18
2. Liver cirrhosis verified by biopsy or appropriate clinic and biochemistry as well as imaging.
3. Written informed consent
4. Speaks and understands Danish

For the subgroup with liver cirrhosis and normal cognition:

1. Normal result in PSE and CRT testing and clinical examination without evidence of HE

   For the subgroup with liver cirrhosis and minimal hepatic encephalopathy:
2. Abnormal result in PSE and / or CRT test, but oriented in time, place and own data.

   For the subgroup with liver cirrhosis and HE grade 2, the following applies:
3. Abnormal PSE and CRT result and / or disoriented in time, place or own data and / or asterixis or other clinical symptoms of HE
4. Ability to collaborate on the performance of CRT test, PSE test and EEG

Inclusion criteria healthy:

1. Liver healthy
2. Age over 18 years
3. Formal education ≤ 14 years
4. Written informed consent
5. Speaks and understands Danish

Inclusion criteria for pre-cirrhosis liver disease:

As for healthy controls plus:

1. In our local outpatient clinic
2. Proven pre-cirrhosis liver disease

Exclusion Criteria:

1. Organic brain disease (eg previous epilepsy, apoplexy, dementia)
2. Hyponatraemia (Na <124 mmol / L)
3. Sepsis one week prior to tests.
4. Heart failure (EC less than 30% or NYHA class III and IV)
5. Severe chronic obstructive pulmonary disease (GOLD stage 3 and 4 ie FEV1 / FVC below 0.7 and FEV1 <50% of expected value)
6. Highly controllable diabetes (HbA1C> 60 mmol / mol)
7. Renal failure (eGFR below 60)
8. Known neurological diseases (epilepsy, stroke, dementia)
9. Intake of coffee or alcohol 6 hours before tests and change of dose in psychoactive drugs within 6 days of the test (morphine, antipsychotics, antidepressants) -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See *cohorts'.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Concordant changes in reaction times and in EEG spectral and frequency analysis | Up to 60 months
  During CRT 150 reaction times are measured. Investigators want to measure if prolonged reaction times >75 percentile are preceded by spectral and frequency changes in EEG. For EEG investigators will assess relative theta and delta activity. EEG and CRT will be done simultaneously.
Observation of cyclic activity in continous reaction times (CRT measures) | Up to 60 months
  Apply mathematically modeled time analysis to establish cyclicity in the 150 measures reaction times and examine if cyclic activity correlates to relative theta and delta activity in the EEG.
Change in EEG spectral and frequency analysis with a clinically indicated standard treatment for minimal hepatic encephalopathy | Up to 60 months
  Some patients will be found eligible for treatment with lactulose or rifaximin due to signs of minimal hepatic encephalopathy. Investigators will use EEG relative theta and delta activity to measure the efficacy of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No
Only anonymized data will be shared if needed due to local regulations.